CLINICAL TRIAL: NCT07254117
Title: The Role of Biochemical and Microbiological Properties of Granulation Tissue in Periodontal Regeneration
Brief Title: The Role of Granulation Tissue in Periodontal Regeneration
Status: Recruiting | Type: Observational
Sponsor: Riga Stradins University (Other)
Collaborators: University of Turku (Other)
Responsible Party: Principal Investigator, Dārta Elizabete Emuliņa, PhD student, Riga Stradins University
Other Study IDs: 2-PĒK-4/434/2025
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Periodontal Bone Loss; Periodontitis; Periodontal Disease; Periodontal Diseases; Periodontal Regeneration; Periodontal Granulation Tissue; Vertical Periodontal Bone Defects; Periodontal Healing
Keywords: Periodontal granulation tissue; Periodontitis; Vertical periodontal bone defects; Vertical defects; Granulation tissue; Periodontal regeneration; Periodontal healing
MeSH Terms: conditions — Alveolar Bone Loss; Periodontitis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Periodontal granulation tissue samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-smoking periodontitis patients: Non-smoking Stage III-IV Grade B-C periodontitis patients with at least one infra-osseous approximal bone defect (with ≥3 mm infrabony component) at premolar-molar region (n=23).
- Smoking periodontitis patients: Smoking Stage III-IV Grade B-C periodontitis patients with at least one infra-osseous approximal bone defect (with ≥3 mm infrabony component) at premolar-molar region (n=23).

SUMMARY:
The goal of this observational study is to distinguish the infectious, healing, and regeneration-related characteristics of two types of gingival granulation tissues, namely infra-osseous and supra-osseous granulation tissues, in people with severe periodontitis (gum disease). Researchers aim to denote if these tissues may play role in healing after periodontal treatment. Researchers will also compare smokers and non-smokers to see if smoking disrupts the healing potential or infectious properties of granulation tissue. Participants will provide gingival fluid (before) and granulation tissue samples (at the time of) periodontal surgery. The main questions this study aims to answer are: 1. Do infra- and supra-osseous granulation tissues have different healing potential and infectious properties? 2. How do these tissues differ in people who smoke compared to people who do not smoke?

DETAILED DESCRIPTION:
This study aims to investigate the biochemical (tissue healing and regenerative) and microbial (infectious) properties of infra- and supra- osseous granulation tissues and compare those characteristics in non-smoking and smoking periodontitis patients. To accomplish these aims, we designed 3 research objectives: 1. To compare the pro-healing and regenerative properties of infra- and supra-osseous granulation tissues harvested from non-smoking periodontitis patients using open-ended proteomics tools. 2. To describe the infectious component of infra- and supra-osseous granulation tissues harvested from non-smoking periodontitis patients using microbiome analysis. 3. To compare the effect of smoking on selected pro-healing, regenerative and virulence markers of infra-osseous granulation tissues. Our main hypothesis is that infra-osseous and supra-osseous granulation tissues of smokers and non-smokers differ from each other in terms of their pro-healing, regenerative and microbial virulence properties, and infra-osseous granulation tissue is a valuable resource for tissue regeneration after periodontal treatment. The demographics of all individuals will be recorded, and full-mouth visible plaque index (PI%), probing pocket depth (PPD), clinical attachment level (CAL) and bleeding on probing (BoP%) scores from six sites of each tooth will be recorded. Periapical radiographs will be taken. Before the surgical applications, all patients will receive full-mouth scaling and root debridement. During the surgical treatment of the residual bone defects, first the supra-osseous granulation tissue samples will be collected. Afterwards, a flap will be raised, and the intra-osseous granulation tissue sample will be collected. Samples will be placed in Eppendorf tubes containing 100 µl of PBS (phosphate buffer saline, pH = 7.2) solution and will be stored at -80°C until laboratory analyses. Proteomics analysis - tissue samples will be homogenized in 100 mM ammonium bicarbonate (ABC) buffer in 2 ml reinforced tubes containing 2.8 mm ceramic (zirconium oxide) beads (Cayman Chemical) using Precellys Bead Mill Homogenizer (Bertin). Microbiome analysis - DNA will be extracted from tissue samples using the DNeasy Blood and Tissue kit following the manufacturer's recommendations (Qiagen, Germany) with minor modifications. Gel electrophoresis using Tapestation 2200 (Genomic DNA and D1000 screentapes, Agilent, USA) will be used to validate product size and purity of a subset of DNA extracts. DNA concentration will be measured using both Nanodrop and Qubit dsDNA BR Assay kit (Thermo Fisher Scientific, USA).

Targeted biochemical analysis - from all tissue samples proinflammatory (IL-1β, IL-6 and TNF-α) and anti-inflammatory (IL-4, IL-10) cytokines, macrophage-activation related chemokines (monocyte chemoattarctant protein C-C motif chemokine ligand 2 (CCL-2/MCP-1), C-C motif chemokine ligand 8 (CCL-8/ MCP-2), C-X-C motif chemokine ligand 9 (CXCL9/MIG), and C-C motif ligand 3 (CCL-3/MIP-1α)), and bone-remodeling marker (osteoprotegerin, Receptor activator of nuclear factor kappa-Β ligand (RANKL), osteocalcin, osteopontin) levels will be measured by Luminex and Simoa techniques, which can detect these markers at levels of femtogram/ml. Luminex 200 bead-based multiplex assay is available at the laboratories of Institute of Dentistry, University of Turku. Simoa HD-X analyzer is available at the laboratories of Turku University Central Hospital. Statistical analysis: Following the detection of the data distribution with the Kolmogorov-Smirnov test, repeated t-test or ANOVA in case of normal distribution will be used in the statistical analysis, and the Mann-Whitney U or Kruskal Wallis tests in case of non-normal distribution. In determining the correlation between healing and virulence marker correlations, the parametric Pearson test or the non-parametric Spearman test will be used according to the distribution. A binary logistic regression analysis with smoking, sex, and age adjustment will be conducted to assess the association between the analytes' levels and the healing response. P < 0.05 will be considered significant. Ethical approval for this project has been received from Riga Stradins University Research Ethics Committee on 28.02.2025. (2-PĒK-4/434/2025). Each patient will be informed about the research objectives and procedures both verbally and through a written informed consent form. They will be notified that, in accordance with patient protection laws, they have the right to withdraw from participation at any time. The patient will also be assured that withdrawing from the study will not affect their future treatment regimen with their periodontologist. Additionally, each patient will be informed that the data obtained during this research will be used to write publications in an anonymous and synthesized manner. All patient visits will be documented, and each patient will be assigned an anonymous patient number. Any necessary corrections to the medical documents will be made by crossing out the incorrect text with a single line and writing the correct text beside it. The clinician will sign next to the correction. If any side effects are observed during the study, the Ethics Committee will be notified.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders.
2. Systemically healthy.
3. Both smokers (smoking at least 10 cigarettes a day or electronic cigarettes daily or quit less than 5 years ago) and non-smokers (never smoked, smoke no more than once a month or quit at least 5 years ago).
4. Patients aged 18 years and over.
5. Patients with a history of severe periodontitis (stage III or IV, grade B-C) and, after completion of the non-surgical stage of periodontal treatment with at least one residual vertical bone defects (with ≥3 mm infrabony component) in premolar-molar region.
6. Patients with a plaque index and bleeding on probing of 20% or lower before surgery.

Exclusion Criteria:

1. Systemic diseases that may affect study results (uncontrolled type 2 diabetes mellitus (HBA1c level of >7%); recent (less than 6 months ago) myocardial infarction or stroke; blood coagulation disorders; recent use of antibiotics (less than 6 months).
2. Use of medications that may affect study results (anti-osteoporotic drugs, statins, corticosteroids, calcium channel blockers, cyclosporine A, antiepileptic drugs, antipsychotic medication or antidepressants, chemotherapy and/or radiotherapy (active or history)).
3. Current pregnancy and/or breastfeeding.
4. Patients who have received any form of systemic antibiotics in the last six months prior to the start of the study.
5. Patients who require antibiotic premedication prior to periodontal treatment.
6. Prosthetic factors in teeth associated with suitable bone defects that prevent clinical measurements.
7. Lack of patient motivation to undertake adequate dental care at home or to complete periodontal treatment.
8. Strong vomiting reflex preventing adequate periodontal treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be formed of two study groups:
  1. Non-smoking Stage III-IV Grade B-C periodontitis patients with at least one infra-osseous approximal bone defect (with ≥3 mm infrabony component) at premolar-molar region (n=23).
  2. Smoking Stage III-IV Grade B-C periodontitis patients with at least one infra-osseous approximal bone defect (with ≥3 mm infrabony component) at premolar-molar region (n=23).
  The sample size for the present cross-sectional study was determined using R (package pwr, function pwr.t.test with type=paired). The effect size, Cohen's D = 0.941, was derived from the Interleukin-10 (IL-10) to total protein ratio. The total sample size was calculated to be 46 patients in two equally sized dependent groups, with a power of 99% (beta = 0.01) and an alpha of 0.05.
  All patients will be recruited from among those enrolled in Riga Stradins University Institute of Stomatology Periodontology Department maintenance treatment program.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of pro-healing/regenerative markers and microbial composition/virulence profiles in infra-osseous and supra-osseous granulation tissues between smokers and non-smokers with Stage III-IV Grade B-C periodontitis. | May 2025 - September 2028
  Regenerative markers: IL-1β, IL-6, TNF-α (pro-inflammatory), IL-4, IL-10 (anti-inflammatory), CCL-2/MCP-1, CCL-8/MCP-2, CXCL9/MIG, CCL-3/MIP-1α (macrophage-activation related chemokines), osteoprotegerin, RANKL, osteocalcin, osteopontin (bone-remodeling markers). Microbial outcomes: presence, abundance, and virulence characteristics of bacteria in infra- and supra-osseous granulation tissue.

SECONDARY OUTCOMES:
Differences in regenerative and microbial markers between infra-osseous and supra-osseous granulation tissues within the non-smoking group. | May 2025 - September 2028
Effect of smoking on selected regenerative and virulence markers in infra-osseous granulation tissue. | May 2025 - September 2028

OTHER OUTCOMES:
Correlation between tissue biochemical/microbial markers and clinical periodontal parameters. | May 2025 - September 2028
  Clinical periodontal parameters, such as probing pocket depth (PPD), clinical attachment level (CAL), bleeding on probing (BoP%), and plaque index (PI%) will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Riga Stradins University Institute of Stomatology, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No